CLINICAL TRIAL: NCT00574119
Title: Effect of Aldosterone on Energy Starvation in Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Marvin W. Kronenberg, M.D., Professor of Medicine and Radiology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB 070824
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-05

CONDITIONS: Heart Failure; Nonischemic Dilated Cardiomyopathy
Keywords: heart failure; positron emission tomography; magnetic resonance imaging; myocardial energetics; myocardial perfusion
MeSH Terms: conditions — Heart Failure | interventions — Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Results with spironolactone (Experimental): patients with heart failure due to nonischemic dilated cardiomyopathy will be studied by 11C acetate positron emission tomography and magnetic resonance imaging using vasodilator and gadolinium to judge myocardial blood flow, before and after 6 months' treatment with spironolactone.
  Interventions: Drug: spironolactone

INTERVENTIONS:
Drug: spironolactone — spironolactone 50 mg daily for 6 months
  Other Names: Aldactone

SUMMARY:
We plan to study the concept of "energy starvation" in heart failure by evaluation of patients with nonischemic dilated cardiomyopathy (NIDCM) (heart failure with reduced heart pump function due to causes other than heart attack). We will use a combination of positron emission tomography and magnetic resonance imaging to study metabolism, anatomy, function, blood flow and efficiency, before and after 6 months' treatment with the drug spironolactone which blocks the deleterious effects of the hormone aldosterone on the myocardium (heart muscle).

DETAILED DESCRIPTION:
Preliminary results showed reduced subendocardial myocardial perfusion reserve in NIDCM compared to normal subjects, and that the degree of impaired perfusion reserve was related to the oxidative metabolic rate as measured by positron emission tomography.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Nonischemic dilated cardiomyopathy
* Left ventricular ejection fraction 35% or less
* Stable heart failure symptoms
* Able to undergo both positron emission tomography and magnetic resonance imaging with gadolinium
* Able to tolerate treatment with spironolactone

Exclusion Criteria:

* Serum potassium >5.0
* Serum creatinine >2.5
* Contraindications to magnetic resonance imaging such as internal cardioverter-defibrillator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marvin W Kronenberg, MD, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Vanderbilt Heart and Vascular Institute, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lawson MA, Hansen DE, Gupta DK, Bell SP, Adkisson DW, Mallugari RR, Sawyer DB, Ooi H, Kronenberg MW. Modification of ventriculo-arterial coupling by spironolactone in nonischemic dilated cardiomyopathy. ESC Heart Fail. 2021 Apr;8(2):1156-1166. doi: 10.1002/ehf2.13161. Epub 2021 Jan 5. PMID 33403831
- [Derived] Bradham WS, Bell SP, Huang S, Harrell FE Jr, Adkisson DW, Lawson MA, Sawyer DB, Ooi H, Kronenberg MW. Timing of Left Ventricular Remodeling in Nonischemic Dilated Cardiomyopathy. Am J Med Sci. 2018 Sep;356(3):262-267. doi: 10.1016/j.amjms.2018.06.003. Epub 2018 Jun 8. PMID 30286821
- [Derived] Lawson MA, Bell SP, Adkisson DW, Wang L, Ooi H, Sawyer DB, Kronenberg MW. High reproducibility of adenosine stress cardiac MR myocardial perfusion imaging in patients with non-ischaemic dilated cardiomyopathy. BMJ Open. 2014 Dec 16;4(12):e005984. doi: 10.1136/bmjopen-2014-005984. PMID 25515841
- [Derived] Bell SP, Adkisson DW, Lawson MA, Wang L, Ooi H, Sawyer DB, Kronenberg MW. Antifailure therapy including spironolactone improves left ventricular energy supply-demand relations in nonischemic dilated cardiomyopathy. J Am Heart Assoc. 2014 Aug 27;3(4):e000883. doi: 10.1161/JAHA.114.000883. PMID 25164945
- [Derived] Bell SP, Adkisson DW, Ooi H, Sawyer DB, Lawson MA, Kronenberg MW. Impairment of subendocardial perfusion reserve and oxidative metabolism in nonischemic dilated cardiomyopathy. J Card Fail. 2013 Dec;19(12):802-10. doi: 10.1016/j.cardfail.2013.10.010. Epub 2013 Oct 29. PMID 24331202

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Results With Spironolactone
Started | 16
Completed | 12
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: one patient excluded prior to drug administration due to normal LV function.
Arm/Group | Results With Spironolactone
Number analyzed (Participants) | 15
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 52 [45 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Work-metabolic Index (WMI) at Baseline
Description: WMI=[left ventricular stroke work/decay rate of 11C-acetate]
Time Frame: baseline
Population: 12 patients completed study
Measure: Median (Inter-Quartile Range); unit: (x10^6), mL x mm Hg/m^2
Arm/Group | Results With Spironolactone
Number analyzed (Participants) | 12
(x10^6), mL x mm Hg/m^2 | 7.4 [2.2 to 3.9]

2. Primary Outcome: Left Ventricular Work-metabolic Index (WMI) at 6 Months
Description: WMI=[left ventricular stroke work/decay rate of 11C-acetate]
Time Frame: 6 months
Population: 12 patients completed study
Measure: Median (Inter-Quartile Range); unit: (x10^6), mL x mm Hg/m^2
Arm/Group | Results With Spironolactone
Number analyzed (Participants) | 12
(x10^6), mL x mm Hg/m^2 | 5.4 [4.4 to 5.9]

3. Primary Outcome: Myocardial Perfusion Reserve Index (MPRI) by Magnetic Resonance Imaging at Baseline
Description: MPRI =calculated myocardial perfusion reserve index based on Gadolinium accretion into myocardium. MPRI was calculated as the ratio of stress/rest relative perfusion upslope, corrected for LV cavity upslope.
Time Frame: baseline
Measure: Mean (Inter-Quartile Range); unit: MPRI
Arm/Group | Results With Spironolactone
Number analyzed (Participants) | 12
MPRI | 1.72 [1.67 to 1.87]

4. Primary Outcome: Myocardial Perfusion Index Reserve (MPRI) by Magnetic Resonance Imaging at 6 Months
Description: as for outcome 3
Time Frame: 6 months
Measure: Mean (Inter-Quartile Range); unit: MPRI
Arm/Group | Results With Spironolactone
Number analyzed (Participants) | 12
MPRI | 1.80 [1.76 to 1.92]

5. Primary Outcome: Change in Myocardial Fibrosis (T1 Time) by Magnetic Resonance Imaging
Description: T1=left ventricular relaxation rate on magnetic resonance imaging, which is correlated with interstitial fibrosis.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Results With Spironolactone
Number analyzed (Participants) | 12
msec | 6 (37)

6. Secondary Outcome: 6 Minute Walk Test (6MWT) at Baseline
Description: 6MWT assesses distance walked over 6 minutes
Time Frame: baseline
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Results With Spironolactone
Number analyzed (Participants) | 12
meters | 521 [468 to 530]

7. Secondary Outcome: 6 Minute Walk Test (6MWT) at 6 Months
Description: 6MWT assesses distance walked over 6 minutes
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Results With Spironolactone
Number analyzed (Participants) | 12
meters | 542 [523 to 604]

8. Secondary Outcome: Minnesota Living With Heart Failure Questionnaire,at Baseline
Description: The questionnaire is comprised of 21 important physical, emotional and socioeconomic ways heart failure can adversely affect a patient's life. Each question is scored from 0 (none or not applicable) to 5 (very much). Total scores range from 0-105. Low scores indicate less adverse impact, while higher scores reflect more adverse impact of heart failure.
Time Frame: baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Results With Spironolactone
Number analyzed (Participants) | 12
score on a scale | 54 [26 to 71]

9. Secondary Outcome: Minnesota Living With Heart Failure Questionnaire.at 6 Months
Description: as for outcome 8
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Results With Spironolactone
Number analyzed (Participants) | 12
score on a scale | 22 [20 to 44]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Results With Spironolactone
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Results With Spironolactone (N=16)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) — shortness of breath during test
pacemaker insertion (Cardiac disorders) | 1 (1) — pacemaker insertion by personal physician

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-02-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT00574119/Prot_SAP_000.pdf